CLINICAL TRIAL: NCT02432677
Title: Evaluation of the Potentiating Effect of Transcranial Direct Current Stimulation (tDCS) on Opioid Analgesia of Pain Threshold in Humans
Brief Title: Evaluation of the Potentiating Effect of tDCS on Opioid Analgesia of Pain Threshold in Humans
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0217
Record Dates: First submitted 2015-04-06; First posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Acute Pain
Keywords: tDCS; Opioid; Pain; Pain threshold
MeSH Terms: conditions — Acute Pain; Pain | interventions — Remifentanil; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Remifentanil + Active tDCS (Experimental): * tDCS session: the procedure will initiate by placing an anode electrode on the primary motor cortex (contralateral to the dominant cortex) and the cathode electrode on the contralateral supra-orbital region. The current employed is 2mA of transcranial direct-current stimulation administered for 20 minutes.
  * Remifentanil - 0,06mcg.kg.min - Infusion 10min before the tDCS session, during the tDCS session and after the tDCS session, until the end of pain tests.
  Interventions: Drug: Remifentanil; Device: Active tDCS
- Placebo + Active tDCS (Other): * tDCS session: the procedure will initiate by placing an anode electrode on the primary motor cortex (contralateral to the dominant cortex) and the cathode electrode on the contralateral supra-orbital region. The current employed is 2mA of transcranial direct-current stimulation administered for 20 minutes.
  * Placebo: Saline infusion - Infusion 10min before the tDCS session, during the tDCS session and after the tDCS session, until the end of pain tests.
  Interventions: Device: Active tDCS; Drug: Placebo
- Remifentanil + Sham tDCS (Other): * Sham tDCS: consists in the same montage of the active tDCS, but the device is turned off 30 seconds after starting stimulation (without letting the patient notice it). The rest of the montage is kept identical to the active one during the 20 minutes session.
  * Remifentanil - 0,06mcg.kg.min - Infusion 10min before the tDCS session, during the tDCS session and after the tDCS session, until the end of pain tests.
  Interventions: Drug: Remifentanil; Device: Sham tDCS
- Placebo + Sham tDCS (Other): * Sham tDCS: consists in the same montage of the active tDCS, but the device is turned off 30 seconds after starting stimulation (without letting the patient notice it). The rest of the montage is kept identical to the active one during the 20 minutes session.
  * Placebo: Saline infusion - Infusion 10min before the tDCS session, during the tDCS session and after the tDCS session, until the end of pain tests.
  Interventions: Device: Sham tDCS; Drug: Placebo

INTERVENTIONS:
Drug: Remifentanil — Remifentanil (IV infusion): 0,06mcg.kg.min. The infusion starts 10min before tDCSThe infusion will be stopped in the event of: a decrease in respiratory rate below 7 breaths / min, a peripheral oxygen saturation below 85%, a lower heart rate of 40 beats per minute, a lower mean arterial pressure of 60 mmHg, sedation causing inadequate management switch stimuli tests and occurrence of vomiting.
  Arms: Remifentanil + Active tDCS; Remifentanil + Sham tDCS
Device: Active tDCS — The stimulation will be administered with a pair of surface electrodes, sponge coated, soaked in saline. A battery-powered constant current stimulator will be used for this purpose (tDCS device). The stimulation is performed by placing the anodal electrode in the primary motor cortex (M1) and the cathodal one in the contralateral supraorbital area and it will use a 2 mA (milliampere) current.
  Other Names: transcranial direct current stimulation
  Arms: Placebo + Active tDCS; Remifentanil + Active tDCS
Device: Sham tDCS — The sham tDCS consists in the same montage of the active tDCS, but the device is turned off 30 seconds after starting stimulation (without letting the patient notice it). The rest of the montage is kept identical to the active one during the 20 minutes session.
  Other Names: Sham - transcranial direct current stimulation
  Arms: Placebo + Sham tDCS; Remifentanil + Sham tDCS
Drug: Placebo — Saline infusion - Infusion 10min before the tDCS session, during the tDCS session and after the tDCS session, until the end of pain tests.
  Arms: Placebo + Active tDCS; Placebo + Sham tDCS

SUMMARY:
The purpose of this study is to evaluate the potential additive effect of tDCS compared to placebo-sham in opioid analgesia on pain thresholds in nociceptive experimental model in healthy volunteers .

DETAILED DESCRIPTION:
Pain is a prevalent symptom in medicine and the role of various opioids is valuable in the treatment of moderate to severe pain. Several technologies of brain stimulation , including transcranial direct current stimulation ( tDCS) are emerging as therapeutic options for many pain conditions. The effect of tDCS was demonstrated in sensory perception , decreasing the threshold for acute pain in healthy volunteers and in various chronic pain conditions . There is evidence about the use of tDCS with the participation through many mechanisms in cortical modulation , including the regulation of neurotransmitters, including opioids. In the context of neurostimulation, opioidergic system and cortical pain modulation, emerge the hypothesis of a possible potentiating effect of tDCS on clinical application of opioid analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Without medication
* Sign the informed consent

Exclusion Criteria:

* Patients who did not understand the Portuguese
* Acute or chronic pain conditions
* Medical or psychiatric disorders
* History of sleep disorders (apnea, hypersomnia, somnambulism…)
* History of alcohol or substance abuse
* Neurological disorder
* Use of anti-inflammatory drugs, steroids and non-steroids, opioid and non-opioid analgesics, psychiatric medications, anticonvulsants, alpha and beta blockers
* Traumatic brain injury
* Neurosurgery
* Metallic implant in the brain

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Thresholds of pain to the cold pressor test (CPT) | 20min

SECONDARY OUTCOMES:
Serum levels of BDNF | 20min
Intensity of electrical brain activity in the bi-spectral index (BIS) | 60min
Sedation level in the visual analogue scale (VAS) | 60min
Temperature of tolerance to the thermal stimulus (TTTS) | 20min
Conditioned pain modulation (CPM) | 20min
  A nociceptive tonic conditioning stimulus - immersion of the non-dominant hand in cold water (0°C for 1 minute) - will be applied concomitant to the progressive thermal stimulus in the dominant forearm as applied in the QST pattern until it reaches the 6/10 pain temperature previously determined by the participant.
Threshold of pain to the thermal stimulus (TT) | 20min
Hemodynamic changes of brain using fNIRSNear-infrared spectroscopy (NIRS) | 60
  The vascular response will be assessed using functional near infrared spectroscopy (fNIRS). Emerging technique that allows the functional mapping of the brain, with a better understanding of the neuro-vascular coupling, the neurophysiological fluctuations and cerebral hemodynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, P.h.D, Principal Investigator — Hospital de Clinicas de Porto Alegre - UFRGS
Locations (1):
- Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Braulio G, Passos SC, Leite F, Schwertner A, Stefani LC, Palmer ACS, Torres ILS, Fregni F, Caumo W. Effects of Transcranial Direct Current Stimulation Block Remifentanil-Induced Hyperalgesia: A Randomized, Double-Blind Clinical Trial. Front Pharmacol. 2018 Feb 19;9:94. doi: 10.3389/fphar.2018.00094. eCollection 2018. PMID 29515438